CLINICAL TRIAL: NCT00965588
Title: A Phase I, Open-Label Study to Evaluate the Safety, Tolerability and Immunogenicity of the UBITh AD Immunotherapeutic Vaccine (UB 311) in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Study to Evaluate Safety, Tolerability and Immunogenicity of Vaccine (UB 311) in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Biomedical (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBI Protocol V118; Protocol V118-AD
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; amyloid beta; vaccine
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (UB 311) (Experimental)
  Interventions: Biological: UB 311

INTERVENTIONS:
Biological: UB 311 — Single liquid dose by intramuscular route at weeks 0, 4, 12.

SUMMARY:
The purpose of this Phase I study is to determine whether the vaccine (UB 311), targeting the amyloid beta peptide (N-terminal amino acids, 1-14), is safe and immunogenic in patients diagnosed with mild or moderate Alzheimer's disease (AD). Amyloid beta was selected as the target antigen based on supporting evidence of the hypothesis that places the accumulation of amyloid beta at the initiating step of AD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate Alzheimer's Disease
* Mini-Mental State Examination (MMSE) 15-25
* Other inclusion criteria apply

Exclusion Criteria:

* Major psychiatric disorder
* Severe systemic disease
* Serious adverse reactions to any vaccine
* Other exclusion criteria apply

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of the vaccine (UB 311). | Screen, treatment & follow-up: 28-30 weeks

SECONDARY OUTCOMES:
To evaluate immunogenicity [and efficacy] of the vaccine (UB 311). | Screen, treatment & follow-up: 28-30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Jang Chiu, M.D., Principal Investigator — National Taiwan University Hospital; Pei-Ning Wang, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital (NTUH), Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Background] Wang CY, Finstad CL, Walfield AM, Sia C, Sokoll KK, Chang TY, Fang XD, Hung CH, Hutter-Paier B, Windisch M. Site-specific UBITh amyloid-beta vaccine for immunotherapy of Alzheimer's disease. Vaccine. 2007 Apr 20;25(16):3041-52. doi: 10.1016/j.vaccine.2007.01.031. Epub 2007 Jan 19. PMID 17287052